CLINICAL TRIAL: NCT06772376
Title: SERS Sensor Based on CHA Reaction for EGFR Mutation Typing in Advanced Lung Cancer: A Multicenter, Open-Label, Double-Blind, Independent Data Analysis Clinical Trial
Brief Title: SERS Sensor Based on CHA Reaction for EGFR Mutation Typing in Advanced Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-045
Record Dates: First submitted 2025-01-03; First posted 2025-01-13 (Actual); Last update posted 2025-03-31 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer in Normal and Malignant Tumors
Keywords: SERS; CHA; EGFR; advanced lung cancer
MeSH Terms: conditions — Neoplasms | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with advanced stage NSCLC by pathology: The study was conducted in 25 centers across the country, recruiting 200 patients with advanced NSCLC with different confirmed EGFR mutation types (Del-19, L858R, T790M, and no gene mutation).
  Interventions: Diagnostic Test: SERS sensor based on CHA reaction

INTERVENTIONS:
Diagnostic Test: SERS sensor based on CHA reaction — 1. Screening interested participants should sign the appropriate informed consent (ICF) prior to completion any study procedures. 2. The investigator will review symptoms, risk factors, and other non-invasive inclusion and exclusion criteria. 3. The following is the general sequence of events during the 3 months evaluation period: 4. Completion of baseline procedures Participants were assessed for 3 months and completed all safety monitoring.
  Other Names: NGS; RT-PCR

SUMMARY:
Summary:This study is a prospective, multicenter clinical study. In previous studies, we successfully constructed a CHA reaction-mediated self-calibrated SERS biosensor for the detection of EGFR mutation typing (Del-19, T790M, L858R) in lung cancer patients, and verified that the accuracy, sensitivity, and specificity of the SERS biosensor exceeded 95% in a small sample of 32 patients. In order to obtain the highest level of clinical evidence and truly achieve clinical transformation, this prospective, multicenter clinical study aims to verify the analytical efficiency of the SERS biosensor for EGFR mutation typing in patients with advanced lung cancer.

Purpose：This prospective, multicenter clinical study aims to verify the analytical efficacy of the previously constructed CHA reaction-mediated self-calibrated SERS biosensor in EGFR mutation typing in patients with advanced lung cancer.

Research subjects: The patients enrolled in this project are confirmed to be advanced non-small cell lung cancer (NSCLC). Enrollment will be completed in 25 centers and the enrollment will be competitive.

Research location: 900th Hospital of Joint Logistics Support Force Research intervention: None Study duration: Patients will be enrolled from June 2024 to June 2025. Subject participation time: Telephone follow-up will be conducted every three months until the end of the study.

DETAILED DESCRIPTION:
With the continuous development of medical technology, especially molecular biology technology, targeted therapy for lung cancer has made rapid progress, and the prognosis of targeted therapy has been significantly improved compared with chemotherapy. In clinical practice, molecular typing of EGFR mutations is conducive to timely and optimal tumor treatment. At present, common detection methods include Sanger sequencing, next-generation sequencing (NGS) and RT-PCR, and most of their samples are from tumor tissues. However, the defects of tissue samples such as small quantity, long detection cycle, heterogeneity and invasiveness have brought challenges to the application of these methods. Therefore, in order to overcome the many limitations faced in detecting gene mutations in tumor tissues, it is of great significance to seek feasible alternatives that are easy to obtain and low intrusiveness for EGFR mutation screening. Previous reports have shown that clinical serum circulating tumor DNA (ctDNA) retains relatively complete genetic information, and EGFR mutations in tumor cells can be reflected in ctDNA in real time. In blood, the detection of ctDNA has unique advantages, such as high timeliness, low false positives and high specificity. Therefore, with blood as an ideal substitute, low-invasive ctDNA detection can become an effective tool for liquid biopsy. Unfortunately, there is no standardized method to detect EGFR mutations in blood samples. Common methods for detecting ctDNA include NGS, mutation amplification retardation system (ARMS) and digital PCR. However, these methods have disadvantages such as complex operation, long time, high cost, low sensitivity and poor specificity. Therefore, a new method for rapid and sensitive ctDNA typing detection is urgently needed.

SERS has become one of the most promising tools in biomedical analysis due to its excellent optical properties. However, since the copy number of mutant ctDNA in blood is only 1% of wild-type DNA, traditional SERS technology cannot meet the strict conditions for ultrasensitive detection. Catalytic hairpin assembly (CHA) is a typical isothermal enzyme-free signal amplification strategy. In order to further improve the analytical ability of the detection platform for low-abundance ctDNA, we combined CHA and SERS as a biosensor constructed as a dual signal amplification strategy to improve the analytical performance of the detection platform for EGFR in serum. In our previous study, we successfully constructed a CHA reaction-mediated self-calibrated SERS biosensor for EGFR mutation typing (Del-19, T790M, L858R) in lung cancer patients, and verified the accuracy, sensitivity, and specificity of the SERS biosensor in a small sample of 32 patients to be over 95%. In order to obtain the highest level of clinical evidence and truly achieve clinical transformation, this prospective, multicenter clinical study aims to verify the analytical efficiency of the SERS biosensor for EGFR mutation typing in advanced lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with Lung cancer meeting the criteria of TNM (Ninth Edition);
2. Participants are willing to participate in this study and follow the research plan;
3. Participants or legally authorized representatives can give written informed consent approved by the Ethics Review Committee that manages the website;

Exclusion Criteria:

1. Patients with other active malignant tumors;
2. Patients with missing baseline clinical data;
3. Patients with severe underlying lung diseases (such as bronchiectasis, bronchial asthma or COPD, etc.), or those with a history of occupational or environmental exposure to dust, mines or asbestos;
4. Participants who do not cooperate or refuse to participate in clinical trials at a later stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with NSCLC by histological pathology and confirmed to be in advanced stage by clinical staging.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
NGS or RT-PCR | through study completion, an average of 1 year
  NGS or RT-PCR for EGFR mutation types
Diagnostic accuracy | through study completion, an average of 1 year
  Determine the EGFR mutation type of cancer patients enrolled through the RAMAN intelligent diagnostic system

SECONDARY OUTCOMES:
SERS(Surface-enhanced Raman spectroscopy) result | through study completion, an average of 1 year
  SERS sensor based on CHA reaction for EGFR mutation types
Time to RAMAN diagnosis | up to 30 days
  The time to perform RAMAN testing and obtain diagnostic results after obtaining serum
Safety assessment Results | up to 30 days
  AEs and SAEs through Day 30